CLINICAL TRIAL: NCT06853782
Title: Comparison of Postoperative Analgesic Efficacy of Transversus Abdominis Plane (TAP) Block and Transversalis Fascia Plane (TFP) Block in Patients Undergoing Elective Total Abdominal Hysterectomy
Brief Title: Comparison of Postoperative Analgesic Efficacy of TAP Block and TFP Block in Patients Undergoing Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, BENSU KARAKOYAK YAĞCI, Anesthesiology and Reanimation Specialist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-22062
Record Dates: First submitted 2025-02-24; First posted 2025-03-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-02

CONDITIONS: Hysterectomy, Benign Uterine Diseases; Abdominal Pain (AP)
Keywords: Transversus Abdominis Plane Block; Transversalis Fascia Plane Block; Total Abdominal Hysterectomy; Postoperative Analgesia; Ultrasound
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP Block Group (Active Comparator): In the TAP block group, the lateral transversus abdominis plane block will be performed by the anesthesiologist under ultrasound guidance using a linear probe after the completion of the surgery. Patients will receive 40 ml of 0.25% bupivacaine, administered in two equal doses, into the fascial plane between the internal oblique muscle and the transversus abdominis muscle on both sides.
  Interventions: Device: High Frequency Linear Probe (GE Logic e R7 Ultrasonography Device, USA)
- TFP Block Group (Active Comparator): In the TFP block group, the transversalis fascia plane block will be performed by the anesthesiologist under ultrasound guidance using a linear probe after the completion of the surgery. Patients will receive 40 ml of 0.25% bupivacaine, administered in two equal doses, between transversus abdominis muscle and transversalis fascia on both sides.
  Interventions: Device: High Frequency Linear Probe (GE Logic e R7 Ultrasonography Device, USA)

INTERVENTIONS:
Device: High Frequency Linear Probe (GE Logic e R7 Ultrasonography Device, USA) — A high frequency linear probe (GE Logic e R7 Ultrasonography Device, USA) device will be used while blocking in both groups.
  Arms: TAP Block Group
Device: High Frequency Linear Probe (GE Logic e R7 Ultrasonography Device, USA) — A high frequency linear probe (GE Logic e R7 Ultrasonography Device, USA) device will be used while blocking in both groups.
  Arms: TFP Block Group

SUMMARY:
Total abdominal hysterectomy is one of the most commonly performed surgeries in women and is known to cause significant pain in especially early postoperative period. The goal of this clinical trial is to compare analgesic efficiacy of TAP block, which is well established by studies in hysterectomy surgeries, and TFP block, a relatively new block with good analgesic effect when used for lower abdominal surgeries, in patients undergoing abdominal hysterectomy surgery.The main parameters to compare the analgesic efficiacy of TAP and TFP blocks are;

1. Pain scores in motion
2. Opioid consumption

Researchers will apply the lateral TAP block and TFP block, prepare the postoperative analgesic treatment regimen and record the patients' analgesic consumption, make ward visits and ask patients about their pain intensity and check for opioid consumption and associated side effects, block-related complications, mobilization, length of hospital stay, and patient satisfaction in patients undergoing elective total abdominal hysterectomy surgery.

Participants will score the pain they feel in motion with certain pain scales.Participants will also respond to the researchers' questions for other parameters in study.

DETAILED DESCRIPTION:
Total abdominal hysterectomy is a commonly performed surgical procedure in women that involves the surgical removal of the uterus and is known to cause significant pain, especially during the early postoperative period.

This study aims to prospectively compare the effects of lateral TAP block and TFP block in patients undergoing elective total abdominal hysterectomy with Pfannenstiel incision under general anesthesia for benign uterine neoplasms in a randomized controlled manner.

The TAP block is a fascial plane block targeting the trunkal T6-T12/L1 nerves located between the internal oblique and transversus abdominis muscles and is an effective regional anesthesia method for abdominal surgeries. In patients undergoing total abdominal hysterectomy, TAP block significantly reduces opioid consumption during the postoperative period and results in marked decreases in pain scores at rest and during movement without causing side effects.

The TFP block is a regional analgesia method used in lower abdominal surgeries targeting the branches of the trunkal T12-L1 nerves, located between the transversus abdominis muscle and transversalis fascia. While the TAP block covers dermatomes from T6-L1, the TFP block targets dermatomes T12-L1. A significant difference from the TAP block is that the TFP block provides effective analgesia in areas innervated by the lateral cutaneous branches emerging from the L1 dermatome that TAP block may not fully cover.

ELIGIBILITY:
Inclusion Criteria:

* ASA scores of 1-2
* Adults aged 18+ years
* Diagnosed with benign uterine neoplasms and will undergo elective total abdominal hysterectomy via Pfannenstiel incision under general anesthesia
* Agreed to participate in the study will be included.

Exclusion Criteria:

* Patients with known

  * Neuropathy
  * Renal failure
  * Hepatic failure
  * Coagulopathy
* Skin infection at the site of intervention
* Allergy to local anesthetics
* BMI > 35 kg/m²
* Hysterectomy surgery extended due to malignancy or multiple surgeries during the same hospitalization
* Emergency surgeries
* ASA scores of 3-4
* Emergency surgery
* Patients who do not consent to participate in the study will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | Postoperative 30th minute, 1st, 2nd, 12th and 24th hours
  Postoperative pain assessment will be performed by a researcher at 30th minutes,1st, 2nd, 12th and 24th hours after the block, using the Numerical Rating Scale (NRS) for pain in movement. Patients will be blinded to the groups they participate in and asked to rate their pain on a scale from 0 to 10, where 0 means no pain and 10 represents the worst pain they can imagine.

SECONDARY OUTCOMES:
Tramadol Consumption | Postoperative 0-6th, 6-12th, 12-24th hours
  Tramadol consumption (between 0-6, 6-12, 12-24 hours) will be assessed by a patient controlled analgesia (PCA) device.
  Additionally, in patients receiving rescue tramadol, the amount of tramadol required will be evaluated by reviewing the patient's daily medication order records.
Rescue Tramadol Need | Postoperative 0-24th hours
  The need for rescue tramadol (Present/Absent), will be assessed by reviewing the patient's daily medication order records.
Adverse Reactions | Postoperative 24th hour
  Opioid associated side effects such as nausea, vomiting, constipation, pruritis, urinary retention, respiratory depression and block related complications will be assessed.
Patient Satisfaction | Postoperative 24th hour
  Patient satisfaction will be assessed by asking patients to choose one of the following options regarding their postoperative comfort: very satisfied, satisfied, neutral, dissatisfied, or very dissatisfied.
Early Mobilization | Postoperative 24th hour
  Early mobilization will be assessed based on whether the patient started to walk within the first 24 hours postoperatively.
Duration of Postoperative Hospital Stay | Postoperative 7th day
  The duration of the postoperative hospital stay will be assessed by checking the operation day and discharge day in the hospital records.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Hospital, Ankara, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Via mail

REFERENCES:
- [Background] Lopez-Gonzalez JM, Lopez-Alvarez S, Jimenez Gomez BM, Arean Gonzalez I, Illodo Miramontes G, Padin Barreiro L. Ultrasound-guided transversalis fascia plane block versus anterior transversus abdominis plane block in outpatient inguinal hernia repair. Rev Esp Anestesiol Reanim. 2016 Nov;63(9):498-504. doi: 10.1016/j.redar.2016.02.005. Epub 2016 Apr 8. English, Spanish. PMID 27067036
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158